CLINICAL TRIAL: NCT06610370
Title: Predicting Postoperative Ambulation Following Selective Dorsal Rhizotomy Based on Preoperative Gross Motor Function Score
Status: Completed | Type: Observational
Sponsor: Acıbadem Atunizade Hospital (Other)
Responsible Party: Principal Investigator, Neslihan Yildizdagi, Physiotherapist, Acıbadem Atunizade Hospital
Other Study IDs: NesliYildizdagi
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Spastic Cerebral Palsy; Walking, Difficulty; Ambulation Difficulty
Keywords: cerebral palsy; ambulation; selective dorsal rhizotomy; gross motor function
MeSH Terms: conditions — Cerebral Palsy; Mobility Limitation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Spastic Cerebral Palsy: 95 children with spastic cerebral palsy were included. Gross Motor Function Measure-88 (GMFM-88) and Gross Motor Function Classification System (GMFCS) were applied to the cases before and after the Selective Dorsal Rhizotomy (SDR) surgery.
  Interventions: Other: Group 1

INTERVENTIONS:
Other: Group 1 — 95 children with spastic cerebral palsy were included. Gross Motor Function Measure-88 (GMFM-88) and Gross Motor Function Classification System (GMFCS) were applied to the cases before and after the Selective Dorsal Rhizotomy (SDR) surgery.

SUMMARY:
Cerebral Palsy (CP) is a neurodevelopmental disorder characterized by abnormalities in muscle tone, movement, and motor skills resulting from permanent, nonprogressive damage to the developing brain before, during, or after birth (Tedla & Reddy, 2021). The worldwide prevalence of CP is 2-3 per 1000 live births (Paul et al., 2022). The most common type of CP is spastic, accounting for approximately 85% of all CP cases (Paul et al., 2022). It is divided into 3 types: hemiparetic, diparetic, and quadriparetic. Selective Dorsal Rhizotomy (SDR) is a surgical technique applied for spasticity management in children with bilateral spastic type CP (Novak et al., 2014). One of the most important points in the decision-making process for SDR surgery is the compatibility of the family's expectations with the expectations of the healthcare professional. Informing the family about the expectations is very important in the decision-making process for surgery (Waite et al., 2023). No study has been found in the literature that provides objective predictive value before surgery in terms of postoperative ambulation. The aim of this study is to examine the predictability of postoperative ambulation status in patients with Spastic Cerebral Palsy (SCP) according to the Gross Motor Function Measure-88 (GMFM-88) score before SDR.

DETAILED DESCRIPTION:
It is an observational study. Purpose of the study: The aim of this study was to examine the predictability of postoperative ambulation status in patients with spastic Cerebral Palsy (SCP) according to the Gross Motor Function Measure-88 (GMFM-88) score before SDR.

95 children with CP were included in the study. Among SCP cases, 71(74.7%) were diparetic, 18(18.9%) were quadriparetic, and 6 (6.3%) were triplegia.

* Can the total score of a gross motor function measure before SDR predict walking after SDR?
* Can the gross motor function measure total score before SDR surgery provide an indication of the family's postoperative walking expectations?

The Gross Motor Function Measure-88 (GMFM-88) and the Gross Motor Function Classification System (GMFCS) were applied to the participants.

ELIGIBILITY:
Inclusion Criteria:

* Age between 0-17,
* Diagnosis of spastic CP,
* Participants and parents willing to participate in the study voluntarily,
* Gross Motor Function Classification System (GMFCS) level between II-IV,
* No history of orthopedic surgery before SDR surgery,
* Actively continuing the Physiotherapy and Rehabilitation (PTR) program for at least 2 months in the post-operative period.

Exclusion Criteria:

* Having different types of CP such as dyskinetic, ataxic and mixed type
* Having hemiparetic type CP
* Having a history of any surgery on the musculoskeletal system before SDR surgery
* Having received Botulinum Toxin injection within the last 6 months.

Ages: 1 Day to 17 Years | Sex: All
Age Groups: Child
Study Population: 95 children with spastic cerebral palsy were included in the study.
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure-88 (GMFM-88) | baseline
  It is an observational scale developed to evaluate gross motor skills and determine limitations in children with CP. Gross motor function is evaluated in 5 sections: supine-prone position and turning, sitting, crawling and kneeling, standing and walking-running and jumping. It consists of a total of 88 items. Each item is scored as 0, 1, 2, 3 or "not tested" and the total score and percentage (%) are calculated.
Gross Motor Function Classification System (GMFCS) | baseline
  It is used to classify motor disorders in children with CP and to describe the severity and course of the disease. The functional status of children with CP is defined in 5 levels. The main difference between the levels is that there is a place for daily living activities. Level I; describes walking without restrictions; level V: describes being carried in a manually propelled wheelchair. The main difference between the levels is that daily life activities also have a place. Every level has its own definition for a variety of ages. The evaluation was made according to the definitions given according to the age of each child.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Altunizade Hospital, Istanbul, AA, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participants data will not be made available to other researchers.